CLINICAL TRIAL: NCT03455803
Title: Effect of CPAP Therapy on Symptoms and Signs of Laryngopharyngeal Reflux Among Patients With Obstructive Sleep Apnea
Brief Title: Effect of CPAP Therapy on LPR Among Patients With OSAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abouelela, Assistant Lecturer, Assiut University
Other Study IDs: 332890
Record Dates: First submitted 2018-02-21; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Laryngopharyngeal Reflux; Obstructive Sleep Apnea
MeSH Terms: conditions — Laryngopharyngeal Reflux; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure

SUMMARY:
This study will investigate the changes in the reflux symptom index (RSI) and reflux finding score (RFS) among patients with obstructive sleep apnea after regular humidified CPAP therapy. Since these two diseases have strong associations then one may consider the possible benefits from therapy in between them.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to stop proton pump inhibitors (PPI) therapy 1 month before enrollment in the study.
* To be eligible as LPR patients in our study, patients must have presented a RSI score > 13 and a RFS score > 7. These thresholds were highly correlated with pathological pH monitoring (pH < 4)

Exclusion Criteria:

* Noncompliance for CPAP Use: According to the standard Medicare criteria to define CPAP compliance, the patients who demonstrated CPAP use ≥ 4 h/ night for ≥ 70% of the nights are considered compliant.
* Antireflux therapy during the period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Reflux symptom index (RSI) change | Change from the baseline RSI at 3 months of regular humidified CPAP application
  Assessment of the changes in the reflux symptom index (RSI) among patients with obstructive sleep apnea according to the determined time frame
Reflux finding score (RFS) change | Change from the baseline RFS at 3 months of regular humidified CPAP application
  Assessment of the changes in the reflux finding score (RFS) among patients with obstructive sleep apnea according to the determined time frame

IPD SHARING:
Plan to Share IPD: No